CLINICAL TRIAL: NCT06363682
Title: Interventional Reference Levels (IRL) in Digestive Endoscopy
Acronym: EndoscopX
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PI225
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-02

CONDITIONS: Each Endoscopic Intervention Using X-rays
Keywords: scopy; X rays; digestive endoscopy; interventional reference levels
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde; Biopsy; Endoscopic Ultrasound-Guided Fine Needle Aspiration; Gastroscopy; Colonoscopy; Dilatation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ERCP — ERCP of the biliary duct ou the pancreatic duct, with or without the use of a stent, in a context of gallstone or tumor or other
  Other Names: ERCP + removal of a biliary stent; ERCP + removal of a pancreatic stent; ECRP + switch of a biliary stent; ERCP + switch of a pancreatic stent; ERCP + cholangioscopy + biopsy; ERCP + clearance of a biliary stent; ERCP + extraction of gallstone; ERCP + placement of a biliary stent; ERCP +placement of a pancreatic stent; ERCP of the pancreatic duct + pancreatoscopy
Procedure: endoscopic ultrasound — The use of endoscopic ultrasound in diverse situation with the necessity of using X rays
  Other Names: endoscopic ultrasound + bulbocholedocian stent; endoscopic ultrasound + hepaticogastric stent; cystogastrostomy with endoscopic ultrasound; endoscopic ultrasound + ponction of a target; endoscopic ultrasound +/- catheterization; endoscopic ultrasound + gastroenterological anastomosis
Procedure: gastroscopy — The diverse procedure in witch scopy is use in orders to place or switch or remove an oesophageal or gastroduodenal stent during a gastroscopy.
  Or for oesophageal or gastroduodenal dilatation.
  Other Names: gastroscopy + removal of gastroduodenal stent; gastroscopy + removal of oesophageal stent; gastroscopy + switch of a oesophageal stent; gastroscopy + placement' of a oesophageal stent; gastroscopy + placement of a gastroduodenal stent; gastroscopy + oesophageal dilatation; gastroscopy + gastroduodenal dilatation
Procedure: Colonoscopy — The diverse procedure in witch scopy is use during a colonoscopy
  Other Names: colonoscopy + placement of a colic stent; colonoscopy + dilatation
Procedure: placement of a nasojejunal tube — placement of a nasojejunal tube for enteral nutritional support

SUMMARY:
Scopy uses X-rays and is not without risk (deterministic and stochastic effects) for the patient and the nursing staff present in the room at the time of an endoscopic procedure requiring its use: its use must be reasoned with a benefit/risk balance in favour of carrying out the interventional procedure. In France, there is currently no multicentre study exploring the radiation doses used for each type of endoscopic procedure.

Main objective: To define IRL (interventional reference levels) adapted to each type of endoscopic procedure.

Secondary objective(s) :

* Application of regulatory texts
* Assessment of patient radiation protection
* Radiation protection assessment for workers

DETAILED DESCRIPTION:
Prospective data collection using an e-CRF available via Easymedstat. Data completed during the endoscopy procedure Completion of a questionnaire by the practitioner who performed the procedure afterwards, including the scopy doses used during the procedure, the type of scopy, the type of intention-to-treat

ELIGIBILITY:
Inclusion Criteria:

* All patients who have received an X-ray dose during an endoscopic procedure

Exclusion Criteria:

* No X-rays produced
* Medical indication not in favour of the scopy procedure in view of the benefit/risk balance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have received an X-ray dose during an endoscopic procedure on one of the 22 private or public hopsitals in France.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-11 (Estimated); Study Completion 2024-06-11 (Estimated)

PRIMARY OUTCOMES:
To define IRL (interventional reference levels) adapted to each type of endoscopic procedure. | From enrollment to the end of data collection at 3 months
  IRL is the mean for all endoscopic procedure using scopy, it is calculated by multiplying the PDS in Gy.cm2 with the time during witch the patient as been expose to Xrays during the procedure

SECONDARY OUTCOMES:
Application of regulatory texts | From enrollment to the end of data collection at 3 months
  yes or no variable : the good delivery of information to the patient about the use of X rays during the procedure ;up-to-date radiation protection training for staff; up-to-date radiation protection training for patient
Assessment of patient radiation protection | From enrollment to the end of data collection at 3 months
  yes or no variable : optimising X-ray doses
Radiation protection assessment for workers | From enrollment to the end of data collection at 3 months
  yes or no variable : Wearing ACTIVE and/or PASSIVE dosimeters in accordance with regulations; Wearing personal protective equipment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University of Nancy, Nancy, Meurthe-et-Moselle, France

IPD SHARING:
Plan to Share IPD: No